CLINICAL TRIAL: NCT05875935
Title: Assessment of Awake Surgery With Electrocorticographic Recordings in the Management of Gliomas and Correlation With Imaging Data
Brief Title: Assessment of Awake Surgery With Electrocorticographic Recordings in the Management of Gliomas and Correlation With Imaging Data (ECoG)
Acronym: ECoG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Medical device defective
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-A02005-52
Record Dates: First submitted 2023-05-04; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Electrocorticography; Karnofski Index; Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject with a non-recurrent glial lesion requiring surgery in vigilance (Experimental)
  Interventions: Procedure: ECoG : electrocorticography

INTERVENTIONS:
Procedure: ECoG : electrocorticography — The skull and the dura are opened under general anesthesia and the two grids of 64 cortical electrodes will be applied to the cortex, one facing the glial lesion, and the other at a distance from the glial lesion in the so-called area. "Healthy" (non-tumor), before the patient wakes up. They consist of 8 recording slides each comprising 8 electrodes of 2 mm in diameter each spaced 0.5 mm (DispoMed®, USA).

SUMMARY:
This study proposes to analyze data from intraoperative ECoG recordings acquired during wakefulness interventions in order to identify the connection networks involved in cognitive functions. This study also proposes to correlate the ECoG data with the imaging data and to analyze the disturbances of the electrophysiological signals induced by the cortical and subcortical brain lesions: this will make it possible to establish a more detailed mapping of the tumor areas and to compare disturbances recorded to those recorded in healthy areas. Thus, this approach should make it possible to improve the quality of excision of glial lesions located in eloquent areas, while reducing the risk of neurological sequelae and thus improve the survival and quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years-old
* Subject with a non-recurrent glial lesion requiring surgery in vigilant condition;
* Brain lesion located in the functional zone;
* Major not protected within the meaning of the law;
* Subject affiliated to a Health Insurance scheme;
* No medical contraindication to performing an MRI (pacemaker);
* No medical contraindication to surgery and anesthesia;
* Karnofski index> 70;
* Subject having signed an informed consent.

Exclusion Criteria:

* Minor subject, pregnant or breastfeeding woman;
* Major subject subject under measure of legal protection, guardianship or deprived of liberty by judicial or administrative decision;
* Subject hospitalized without consent;
* Subject treated with antipsychotics (neuroleptic or lithium);
* Subject who has already been treated for his glial lesion by surgery and / or radiotherapy;
* Subject refusing to sign an informed consent.
* Subject wishing to discontinue participation in the study before completion;
* Subject for which the surgical intervention and / or the ECoG recording could not be carried out after admission to the operating room (whatever the reason).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
electrocorticographic recordings | 12 months
  Intraoperative ECoG recordings (raw signals) acquired during awake surgery which in clinical practice couples cortical stimulation and simultaneous ECoG recordings with behavioral tests. The regions defined as electrophysiologically "connected" to the stimulated region will be those for which an afterdischarge is recorded (short-duration rhythmic activity following the stimulation) and/or a cortico-cortical evoked potential is obtained after a average of 5 successive stimulations.

CONTACTS AND LOCATIONS:
Locations (1):
- Clairval Private Hospital, Marseille, Paca, France